CLINICAL TRIAL: NCT00738621
Title: A Comparison of Combination Antiemetic Regimen for Prevention of PONV in Breast Surgery Patients
Brief Title: Combination Antiemetic Regimen for Prevention of PONV in Breast Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Richard Beswick, Scott and White Healthcare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Scott and White
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2008-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; breast surgery; prevention; antiemetics
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral aprepitant 40 mg - given within 3 hours prior to induction dexamethasone (4mg intravenous) administered immediately after induction ondansetron (4mg (2ml) intravenous) administered at cessation of anesthesia
  Interventions: Drug: Aprepitant, Dexamethasone, Ondansetron
- A,2 (Placebo Comparator): Oral aprepitant 40 mg- given within 3 hours prior to induction dexamethasone (4mg intravenous) administered immediately after induction Placebo ( intravenous saline 2ml) administered at cessation of anesthesia
  Interventions: Drug: Aprepitant, Dexamethasone, Placebo

INTERVENTIONS:
Drug: Aprepitant, Dexamethasone, Ondansetron — Aprepitant oral 40mg one dose, dexamethasone IV 4mg one dose, ondansetron 4 mg one dose
  Other Names: Emend=aprepitant
  Arms: 1
Drug: Aprepitant, Dexamethasone, Placebo — Aprepitant 40mg oral one time, dexamethasone IV 4mg one time placebo one time
  Other Names: Emend=aprepitant
  Arms: A,2

SUMMARY:
The purpose of this study is to compare the efficacy of the use of oral aprepitant in combination with intravenous ondansetron and dexamethasone with the efficacy provided by the use of oral aprepitant and dexamethasone for preventing vomiting during the first 24-48 hours after breast surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is one of the most common complications associated with surgery. The overall incidence of PONV is reported to be about 25-30% with specific surgeries having an incidence up to 70-80%.1-5 Although PONV is typically not life threatening, patients dread the sensation of nausea and the serious effects of retching and vomiting. PONV in the surgical patient can cause wound dehiscence, electrolyte imbalance, increased intraocular pressure, increased intracranial pressure, aspiration, esophageal rupture, and loss of vision due to retinal detachment. 6-11 In several studies, investigators found that patients rank vomiting as the most undesirable common side effect after surgery. PONV is costly in economic terms and is a reason day surgery patients must be admitted in the hospital for an overnight stay.12, 13 It is estimated that a patient who experiences an episode of vomiting costs an additional $300 based on emesis basins, supplies, gowns, bedding, additional medications, and nursing/physician time.14-20

In general, PONV is highest in women (with a 2-3 times increased risk) and particularly after procedures such as gynecological surgery, laparoscopy, thyroidectomy and breast surgery.5, 21-35 A study by Sinclair and group found that patients undergoing breast augmentation experienced an 8-10 fold higher incidence of PONV than patients undergoing other types of plastic surgery.26 Similar incidences were found in other studies of 48% to 68% of PONV in patients undergoing mastectomies, breast reconstruction, and implantation.36-40

The hospitalization of patients undergoing breast cancer surgery has significantly decreased by 40% between 1993 and 2003. Many surgeries are now being performed on an outpatient basis according to the Agency for Healthcare Research and Quality (AHRQ), with 96% of lumpectomies, 86% of partial mastectomies and 22% of complete mastectomies scheduled as ambulatory surgeries.41 Carroll and group found that 35% of outpatients suffered from nausea and vomiting after they left the surgical center.42 Therefore, the resulting problem is not only the high incidence of nausea and vomiting in this specific group of patients but the post discharge nausea and vomiting (PDNV) that will occur when these patients are at home and without direct medical oversight.

Although still unclear, it is postulated that the etiology of postoperative nausea and vomiting is the central mechanism involving stimulation of the chemoreceptor trigger zone (CTZ) located bilaterally at the floor of the fourth ventricle in the area postrema. The CTZ is sensitive to toxins and other substances in the blood and cerebrospinal fluid. The CTZ also receives sensory signals from the gastro-intestinal tract. The are three major central nervous system (CNS) areas involved with PONV which all have specific emetogenic receptors. Blockade of these receptors is postulated to be the mechanism of action of the commonly used antiemetics. The agents' antagonist activity may be at one or more receptors with different binding affinities and acting at different emetic neuroreceptors. The multifactorial etiology of PONV involving multiple receptors is believed to be the reason one single agent is not 100% effective. The administration of an agent working on one receptor type will typically reduce the PONV incidence by 30%. Use of a combination of antiemetic agents acting on different receptor sites will further reduce the incidence. This combination has shown greater efficacy than a single agent alone. Although this regimen has improved outcomes it has not eliminated the problem of PONV and patients needing rescue therapy post surgery occurs frequently. It would appear reasonable to assume that the use of more than 2 antiemetics would further reduce the incidence of PONV.43 However; published evidence of greater than 2 agents is scarce. Therefore, the main objective of our proposal is to study a combination antiemetic regimen (3 agents vs. 2 agents) in females scheduled for breast surgery, a patient population considered at high risk for postoperative vomiting. The selected agents will cover different receptors based on the hypothesized PONV multifactorial etiology with stimulation of several factors. It is unknown which of these receptors may be stimulated and by which stimuli (anesthetic, surgery, or patient factors).

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met for the potential subject to be eligible for participation:

1. The subject is a female scheduled to undergo ambulatory breast surgery performed under general anesthesia
2. The subject is expected to undergo general inhalation anesthesia.
3. The subject presents with two of the three following high-risk factors associated with PONV (must be in their medical history in order to be eligible)

   * She is a non-smoker.
   * She has documented history of PONV and/or motion sickness.
   * She is expected to receive intra-operative and postoperative opioid.
4. The subject's American Society of Anesthesiologist physical status is ASA I-III
5. The subject is between18 to 65 years of age.
6. The subject is expected to be discharged from the hospital/surgical center on the same day as the surgery.
7. The subject has provided written informed consent to participate in the study.

If any of the following exclusion criteria are met, the potential subject is NOT eligible for participation:

1. The subject has a history of allergic reaction to, intolerances of or contraindications for any of the study medications or required anesthetic agents.
2. The subject has received or is expected to receive any excluded preoperative drug within 48 hours prior to induction; or is expected to receive any excluded intra-operative or postoperative medications.
3. The subject is pregnant or lactating. (If the potential subject is pre-menopausal, a urine pregnancy test must be performed within 24 hours/1 day of study prior to the planned surgery time and confirmed negative in order for the potential subject to be enrolled).
4. The subject is taking warfarin.
5. The subject has a history of alcohol and/or drug abuse within 1 year of study medication, or has a positive screening or pre-study test for alcohol or drugs of abuse.
6. The subject is expected to require the use of a nasogastric tube postoperatively.
7. The subject has a diagnosed latex allergy.
8. The subject has used oral aprepitant (Emend®) within the last 30 days.
9. The subject has participated in a randomized study or has been exposed to any experimental drug within 30 days prior to enrollment of this study.

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of the use of oral aprepitant in combination with intravenous ondansetron and dexamethasone with the efficacy provided by the use of oral aprepitant in combination with dexamethasone alone for preventing vomiting for 1st 24hrs | 2 yrs

SECONDARY OUTCOMES:
Compare efficacy of oral aprepitant in combination with IV ondansetron and dexamethasone with efficacy of dexamethasone and oral aprepitant alone for preventing vomiting during the 24-48 hours after breast surgery | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Tricia A Meyer, PharmD, Principal Investigator — Scott and White Healthcare
Locations (1):
- Scott and White Healthcare, Temple, Texas, United States